CLINICAL TRIAL: NCT01497626
Title: A Phase I Study of the HER1, HER2 Dual Kinase Inhibitor, Lapatinib Plus the Proteosomal Inhibitor Bortezomib in Patients With Advanced Malignancies
Brief Title: Lapatinib and Bortezomib in Patients With Advanced Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug support withdrawn
Sponsor: Georgetown University (Other)
Collaborators: GlaxoSmithKline (Industry); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-533; XO5371 (Other: Millennium Pharmaceuticals); 8LAP114999 (Other: GlaxoSmithKline)
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2015-09

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced cancer; Solid tumor
MeSH Terms: interventions — Lapatinib; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib plus lapatinib (Experimental): Combination treatment with lapatinib and bortezomib
  Interventions: Drug: Lapatinib and bortezomib

INTERVENTIONS:
Drug: Lapatinib and bortezomib — Lapatinib will be taken orally continuously for 28 days of each 28-day cycle, including a run-in of lapatinib alone day -7 to day 1 of cycle 1.
  Bortezomib will be administered IV on days 1, 8, and 15 of each cycle. The exact doses of both drugs will be dependent on which cohort the subject is in and adverse events observed in previous cohorts.
  Other Names: Velcade

SUMMARY:
This study is for patients with an advanced type of cancer for which no curative treatment exists.

The purpose of this study is to test the safety and efficacy of the combination of the study drugs, lapatinib and bortezomib. Lapatinib is a drug that targets two proteins important for the growth of cancer cells known as HER1 (EGFR) and HER2. By inhibiting these proteins, lapatinib can inhibit cancer cell growth and even lead to their death. Lapatinib is an oral pill given by mouth once every day. Lapatinib is approved by the FDA for patients with breast cancer.

Bortezomib is a drug that targets a part of cancer cells known as the proteosome. By inhibiting the proteosome, bortezomib can inhibit cancer cell growth and even lead to their death. Bortezomib is given intravenously, once a week, 2 out of every 3 weeks. Bortezomib is approved by the FDA for patients with multiple myeloma and mantle cell lymphoma.

This research is being done because it is not known if the combination of lapatinib and bortezomib will work better than lapatinib or bortezomib alone, although in the lab and in animal studies the combination of the two drugs was much more effective than either drug alone.

As part of this study biopsies will be taken of patients' tumors before any treatment, after starting lapatinib alone, and after receiving both lapatinib and bortezomib. Investigators want to study what markers inside tumors may relate to how well these two medications work. These biopsies are required as part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven malignant solid tumor with measurable disease
* Progression on, or intolerance of, or ineligibility for all standard therapies
* Biopsy accessible tumor deposits
* LVEF >/= institutional normal
* Corrected QT interval less than 500 milliseconds by EKG
* ECOG performance status 0-2
* Subjects with no brain metastases or a history of previously treated brain metastases who have been treated by surgery or stereotactic radiosurgery at least 4 weeks prior to enrollment and have a baseline MRI that shows no evidence of active intercranial disease and have not had treatment with steroids within 1 week of enrollment.
* Adequate hepatic, bone marrow, and renal function
* Partial thromboplastin time must be </= 1.5 x upper limit of institution's normal range and INR < 1.5. Subjects on anticoagulants will be permitted to enroll as long as the INR is in the acceptable therapeutic range.
* Life expectancy > 12 weeks
* Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to initiation of treatment and/or postmenopausal women must be amenorrheic for at least 12 months.
* Subject is capable of understanding and complying with parameters as outlines in the protocol and able to sign and date the informed consent form.

Exclusion Criteria:

* Patients with lymphomas
* CNS metastases which do not meet the criteria outlines in the inclusion criteria
* Peripheral neuropathy >/= Grade 2 at baseline or peripheral neuropathy >/= Grade 1 with neuropathic pain
* Active severe infection or known chronic infection with HIV or hepatitis B virus
* Cardiovascular disease problems including unstable angina, therapy for life-threatening ventricular arrhythmia, or myocardial infarction, stroke, or congestive heart failure within the last 6 months
* Life-threatening visceral disease or other severe concurrent disease
* Women who are pregnant or breastfeeding
* Anticipated patient survival under 3 months
* Concurrent use of known CYP 3A4 inhibiting or activating medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 18 months
  The highest dose at which </= 1 out of 6 subjects has a dose-limiting toxicity

SECONDARY OUTCOMES:
toxicity | 18 months
  Adverse events seen during the trial graded using CTCAE version 4
Response rate | 18 months
  complete response and partial response measured by RECIST 1.1
Disease control rate | 2 months
  stable disease after two cycles+ partial response + complete response as determined by RECIST 1.1 criteria
Pharmacodynamics | pre-treatment, after 1 week of therapy and adter 3 weeks of therapy
  To assess changes in the following in serial tumor samples: EGFR, HER2, HER3, AKT, Actin, ERK, GSK3a-beta, IGF-1R, MEK 1/2, mTOR, p70S6, P13K, PTEN, SHC Y317, NFKB, IKB, CFK4, CDK2, cyclin D1, cyclin A, Cyclin E, p15, p16, p21, p27, beta-catenin, and ras gene mutation

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pishvaian, MD PhD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Lynce F, Wang H, Petricoin EF, Pohlmann PR, Smaglo B, Hwang J, He AR, Subramaniam DS, Deeken J, Marshall J, Pishvaian MJ. A phase I study of HER1, HER2 dual kinase inhibitor lapatinib plus the proteasome inhibitor bortezomib in patients with advanced malignancies. Cancer Chemother Pharmacol. 2019 Nov;84(5):1145-1151. doi: 10.1007/s00280-019-03947-7. Epub 2019 Sep 19. PMID 31538230